CLINICAL TRIAL: NCT05234931
Title: Traumatic Anal Sphincteric Injury Immediate vs Delayed Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Youssef Mohamed Ali, DOCTOR, Assiut University
Other Study IDs: anal sphincteric injury
Record Dates: First submitted 2022-01-30; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Traumatic Anal Sphincteric Injury,Immediate vs Delayed Repair

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
comparison between immediate and delayed repair regarding the need for another technique ,pain score or repositioning and need for repair. We aim to evaluate the effects of immediate and delayed repair regarding the morbidity and mortalit

* Objective 1: to assess the operative time and surgical field of both choices.
* Objective 2: to estimate post-operative pain using pain score, to measure hospital stay and to assess short -term post-operative complications

DETAILED DESCRIPTION:
Many different secondary procedures have been described in an attempt to restore continence. These may be classified into indirect methods, where the divided sphincter is left unrepaired, and direct methods to repair the sphincter itself. Indirect techniques include construction of circum anal slings of striated muscle or fascia external sphincter reefing procedures" and the use of striated muscle grafts. Direct methods involve identification, mobilization, and suture of the ends of the divided sphincter. Thearliest 'attempts employed an end-to-end

ELIGIBILITY:
Inclusion Criteria:

1. both sex
2. - Traumatic Patients Who Presented by anal Sphincteric Injury
3. accept to participate in the study

Exclusion Criteria:

1. Patient who arrest immediately when arrived trauma unit
2. Obstetric Patients Who Presented by anal Sphincteric Injury

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: sample size was calculated using epidemiological information statistical package version7 Based on paramaters for cross sectional study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
comparison between immediate and delayed repair | Baseline
  Regarding the need for another technique ,pain score or repositioning and need for repair. We aim to evaluate the effects of immediate and delayed repair regarding the morbidity and mortalit
  * Objective 1: to assess the operative time and surgical field of both choices.
  * Objective 2: to estimate post-operative pain using pain score, to measure hospital stay and to assess short -term post-operative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Result] Koscinski T, Marti MC. [Treatment of fecal incontinence by overlapping sphincteroplasty]. Wiad Lek. 1997;50 Suppl 1 Pt 1:151-4. Polish. PMID 9446343
- [Result] Barisic G, Krivokapic Z, Markovic V, Popovic M, Saranovic D, Marsavelska A. The role of overlapping sphincteroplasty in traumatic fecal incontinence. Acta Chir Iugosl. 2000;47(4 Suppl 1):37-41. PMID 11432241
- [Result] KRAATZ H. [PLASTIC SURGERY OF THE SPHINCTER FOR THE CONTROL OF INCONTINENCE]. Acta Chir Acad Sci Hung. 1964;5:219-23. No abstract available. German. PMID 14230622